CLINICAL TRIAL: NCT01832649
Title: Effectiveness of an Exercise Program in the Treatment of Cocaine Dependence
Brief Title: Exercise as an Adjunctive Treatment for Cocaine Dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-PEF-2011-98
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Cocaine Dependence
Keywords: Exercise; Cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Moderate-vigorous intensity strength exercise. 50 minutes per session, 2 times per week, 8 weeks.
  Interventions: Behavioral: Exercise
- Health education (Active Comparator): Health education sessions. 50 minutes per session, 2 times per week, 8 weeks.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Exercise — Supervised moderate-vigorous exercise in group, based on strength and calisthenics exercises, 2 times per week during 8 weeks.
  Arms: Exercise
Behavioral: Health education — Supervised groups 2 times per week during 8 weeks.
  Arms: Health education

SUMMARY:
The purpose of this study is to evaluate if exercise added to usual treatment improves cocaine dependence treatment. The primary objective of this study is to investigate if exercise can facilitate cocaine craving reduction. The secondary aims are to evaluate if exercise can reduce negative mood states, improve quality of life and facilitate abstinence of cocaine.

DETAILED DESCRIPTION:
This study is designed as two-groups, randomized controlled trial to evaluate the effectiveness of an 8-week exercise program added to usual treatment compared with a health education program in 20 cocaine dependent patients. These participants will be randomized to one of the following two groups: a) exercise group: supervised moderate-vigorous exercise in group based on strength and calisthenics exercises, b) control group: supervised health education in group. All participants must have DSM-IV diagnosis of cocaine dependence as the primary disorder and must be in treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of cocaine dependence as primary disorder
* age between 18 and 60 years
* current psychosocial cocaine treatment

Exclusion Criteria:

* medical problems that contraindicate the participation in an exercise program
* family history of sudden death and/or early death due to cardiovascular reasons
* current inclusion in a regular exercise program

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cocaine craving measured by means of a 5-item craving questionnaire (Roger D. Weiss) | weekly, up to 8 weeks

SECONDARY OUTCOMES:
Mood states measured by Profile of Mood States (POMS) | weekly, up to 8 weeks
Quality of life measured by 36-item Short-Form Survey (SF-36) | monthly, up to 2 months
Change in Physical fitness (BMI, functional capacity and strength) | Change from Baseline Physical Fitness at 2 months
Percent days abstinent defined as the ratio between the number of negative cocaine urine test and the number of realised cocaine urine test | weekly, up to 8 weeks
Change in cocaine craving measured by means of visual analogue scale (VAS) | Change from Baseline Cocaine Craving at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Siñol Llosa, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain